CLINICAL TRIAL: NCT03061604
Title: A Randomized Control Study to Determine the Efficacy and Safety of Combining Hemospray With Medical Standard of Care Treatment in the Management of Acute Variceal Bleeding in Cirrhotic Patients.
Brief Title: RCT to Determine the Efficacy of Combining Hemospray With Medical Treatment in Acute Variceal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Mostafa Ibrahim, Principal Investigator, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hemospray Varices RCT
Record Dates: First submitted 2016-11-30; First posted 2017-02-23 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Variceal Hemorrhage
MeSH Terms: interventions — Octreotide; Blood Transfusion; Ceftriaxone; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemospray (Experimental): All subjects will be treated by medical treatment in the terms of combination of vasoactive medication, blood transfusion and Ceftriaxone PLUS Hemospray treatment within 2 hours of admission.
  The medical treatment will be continued till 12 hours after admission and then second endoscopy will be performed (12-24 hours after admission).
  Interventions: Device: Hemospray; Drug: Octreotide; Biological: Blood transfusion; Drug: Ceftriaxone
- Non Hemospray (Active Comparator): All subjects will be treated by medical treatment in the terms of combination of Octreotide, blood transfusion and Ceftriaxone.
  The medical treatment will be continued till 12 hours after admission and then second endoscopy will be performed (12-24 hours after admission).
  Interventions: Drug: Octreotide; Biological: Blood transfusion; Drug: Ceftriaxone

INTERVENTIONS:
Device: Hemospray — Hemospray is a novel hemostatic powder licensed for endoscopic hemostasis of non-variceal upper gastrointestinal bleeding which has been shown to be effective in preliminary studies for the management of patients with peptic ulcer bleeding, including those on anticoagulant or antithrombotic therapy . Recently, two case reports and a pilot study reported that hemostatic powder may be useful in emergency management of variceal bleeding as a bridge towards more definitive therapy
  Other Names: Hemostatic Powder
  Arms: Hemospray
Drug: Octreotide — Octreotide will be administered to all patients at time of admission and will be continued for 24 hours
  • Dosage: 50 mcg bolus at admission then 25 mcg/hour
  Other Names: Vasoactive drug
Biological: Blood transfusion — Blood transfusion will be administered to all patients if needed
Drug: Ceftriaxone — Ceftriaxone will be administered to all patients on daily basis
  Other Names: Antibiotics

SUMMARY:
INTRODUCTION Acute variceal bleeding (AVB) is a severe complication of portal hypertension in patients with liver cirrhosis. The primary therapy includes the administration of vasoactive drugs, antibiotics and endoscopic therapy; preferably esophageal banding ligation (EBL) and/or cyanoacrylate injection when bleeding occurs from gastric varices.

In this context, the idea is to assess "Hemospray" (Cook Medical, Winston-Salem, NC) as an initial therapy in patients with massive bleeding as a temporary "bridge" until definitive treatment could be instituted.

The data generated from the pilot study performed between Erasme hospital, ULB and TBRI , Cairo showed that adding Hemospray as early as possible in the management steps could increase the bleeding control rate up to 95 % at 24 hours.

OBJECTIVE The primary efficacy objective of this study is to assess the efficacy of Hemospray in combination with standard of care (SOC) medical treatment compared to the efficacy of SOC in the Control Arm in patient with acute variceal bleeding in cirrhotic patient.

The primary safety objective of this study is to evaluate the safety of Hemospray when used in combination with SOC compared to SOC in the Control Arm.

1.1. Secondary:

* To evaluate the effect of timing of Hemospray treatment on the outcomes of bleeding patients
* To evaluate the adverse effects on both therapeutic regimens (SAEs and clinically significant AEs).

DETAILED DESCRIPTION:
STUDY ENDPOINTS :

1.1. Primary endpoint: Hemostasis is the primary end point: which is a combined endpoint of Endoscopic hemostasis at (12-24) hours and Clinical hemostasis during (12-24) hours.

1.2. Secondary endpoints:

* Need for rescue endoscopy (Before 12h)
* Safety
* Interaction with coagulation profile
* Rebleeding at 5 days.
* Survival at 5 days
* Survival at 30 days

ELIGIBILITY:
Inclusion Criteria:

* Subject must be over 18 years of age.
* Suspected or proven acute variceal bleeding , Gastric lavage will be done for all patients at admission (Acute bleeding is confirmed on the presence of blood in stomach)
* Subjects must be willing to give written informed consent for the trial
* Known or suspected cirrhosis

Exclusion Criteria:

* Patient is: < 18 years of age
* Unable to consent
* Contraindicated to undergo endoscopy,
* Already hospitalized for another illness
* Pregnant or lactating
* Patients with altered post-surgical anatomy of the stomach
* Previously placed intrahepatic portosystemic shunt
* Patient treated by other endoscopic or surgical modalities within 30 days prior to the intended application of Hemospray

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Haemostasis | 24 hours
  which is a combined endpoint of Endoscopic hemostasis at (12-24) hours and Clinical hemostasis during (12-24) hours.

SECONDARY OUTCOMES:
Need for rescue endoscopy | 12 hours
Survival | 5 days
Survival | 15 days
Survival | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Deviere, PHD, Study Director — Erasme Hospital , Université libre de Bruxelles
Locations (2):
- Erasme Hospital , ULB, Brussels, Belgium
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
If data will be shared to other researchers , The patients personal data will be removed

REFERENCES:
- [Derived] Ibrahim M, El-Mikkawy A, Abdel Hamid M, Abdalla H, Lemmers A, Mostafa I, Deviere J. Early application of haemostatic powder added to standard management for oesophagogastric variceal bleeding: a randomised trial. Gut. 2019 May;68(5):844-853. doi: 10.1136/gutjnl-2017-314653. Epub 2018 May 5. PMID 29730601